CLINICAL TRIAL: NCT04336332
Title: Randomized Comparison of Combination Azithromycin and Hydroxychloroquine vs. Hydroxychloroquine Alone for the Treatment of Confirmed COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Ineffectiveness of treatment
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Sabiha Hussain, MD,MPH, Associate Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 002011; Pro2020000712 (Other: Rutgers Health Sciences IRB); Pro2020000712 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Hydroxychloroquine Sulfate + Azithromycin (Experimental): * Hydroxychloroquine sulfate 200 mg taken by mouth three (3) times a day for 10 days
  * Azithromycin 500 mg taken by mouth on Day 1, followed by
  * Azithromycin 250 mg taken by mouth once (1) time a day for four (4) days.
  Interventions: Combination Product: Hydroxychloroquine Sulfate + Azithromycin; Drug: Hydroxychloroquine Sulfate
- Arm 2: Hydroxychloroquine Sulfate alone (Experimental): • Hydroxychloroquine sulfate 200 mg taken by mouth three (3) times a day for 10 days
  Interventions: Drug: Hydroxychloroquine Sulfate
- Arm 3: Placebo (No Intervention): * Placebo pills Days 1-6.
  * If you still have COVID-19 symptoms you will receive Hydroxychloroquine sulfate 200 mg by mouth three (3) times a day for 10 days

INTERVENTIONS:
Combination Product: Hydroxychloroquine Sulfate + Azithromycin — Given PO
  Other Names: Hydroxychloroquine; Plaquenil; Z-Pak; Zithromax; Zmax
  Arms: Arm 1: Hydroxychloroquine Sulfate + Azithromycin
Drug: Hydroxychloroquine Sulfate — Given PO
  Other Names: Hydroxychloroquine; Plaquenil
  Arms: Arm 1: Hydroxychloroquine Sulfate + Azithromycin; Arm 2: Hydroxychloroquine Sulfate alone

SUMMARY:
This is a three-arm randomized trial comparing the efficacy of single agent hydroxychloroquine to the combination of hydroxychloroquine and azithromycin, and to a delayed hydroxychloroquine regimen, which will serve as a contemporaneous Day 1-6 supportive care control, in eliminating detectable SARS-CoV-2 on day 6 following the initiation of treatment in order to determine which regimen is more effective.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine change in viral load at day 6 compared to baseline between two regimens to treat COVID-19 and a contemporaneous control group.

SECONDARY OBJECTIVES:

I. Time to resolution of symptoms (symptom questionnaire)

II. Change in the fever curve resulting in shorter time to afebrile for 48 hours

III. Normalization of vital signs

IV. Time to discharge (if hospitalized)

V. Assessment of agent toxicity as measured by standard metrics

VI. Collection of throat swab and blood for viral load, presence of IgM or IgG antibodies

VII. If feasible on samples collected for quantitative PCR decrease in virus shedding (in oropharyngeal secretions)

VIII. Measures of cytokines in blood including IL6, IL-8, TNF, INF

IX. Routine standard of care labs obtained as part of the care of these patients such as differential white count, CRP, troponin and LFTs will be analyzed for correlative trends

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven SARS-CoV-2 infection by an accepted assay with symptoms consistent with COVID-19
* Ability to measure and quantify viral load by quantitative PCR
* Age 18 to 89
* Ability to swallow oral medications
* Patients must read, understand and sign IRB approved informed consent

Exclusion Criteria:

* Pregnancy or women who are breast feeding
* Two consecutive negative assays for SARS-CoV-2 infection
* Patients that lack decision-making capacity will not be approached to participate in this study
* Inability to tolerate oral medications
* Allergy or prior adverse reaction to either azithromycin or hydroxychloroquine sulfate
* QTc interval > 470 mSEC
* History of ongoing ventricular cardiac dysrhythmias of grade 2 as described by NCI CTCAE 5.0 criteria
* History of serious ventricular arrhythmia (VT or VF > 3 beats in a row)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Hussain, MD, Principal Investigator — Rutgers, The State University of New Jersey; Steven K. Libutti, MD, FACS, Study Chair — Rutgers Cancer Institute of New Jersey
Locations (5):
- United States (5):
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Robert Wood Johnson University Hopsital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The University Hospital, Newark, New Jersey
  - University Hospital-Newark, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Hydroxychloroquine Sulfate + Azithromycin: * Hydroxychloroquine sulfate 200 mg taken by mouth three (3) times a day for 10 days
  * Azithromycin 500 mg taken by mouth on Day 1, followed by
  * Azithromycin 250 mg taken by mouth once (1) time a day for four (4) days.
  Hydroxychloroquine Sulfate + Azithromycin: Given PO
  Hydroxychloroquine Sulfate: Given PO
Period: Overall Study
Arm/Group | Arm 1: Hydroxychloroquine Sulfate + Azithromycin | Arm 2: Hydroxychloroquine Sulfate Alone | Arm 3: Placebo
Started | 16 | 30 | 29
Completed | 16 | 30 | 29
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Hydroxychloroquine Sulfate + Azithromycin | Arm 2: Hydroxychloroquine Sulfate Alone | Arm 3: Placebo | Total
Number analyzed (Participants) | 16 | 30 | 29 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 11 | 19 | 18 | 48
  >=65 years | 5 | 10 | 11 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 12 | 29
  Male | 9 | 20 | 17 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 7 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 2 | 4 | 6
  White | 12 | 15 | 20 | 47
  More than one race | 2 | 5 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 30 | 29 | 75

OUTCOME MEASURES:

1. Primary Outcome: Changes in Patients Viral Load
Description: Will be assessed at day six compared to baseline between hydroxychloroquine sulfate alone and hydroxychloroquine sulfate plus azithromycin to treat COVID-19.
Time Frame: Baseline and day six
Population: Data were not collected
Arm/Group | Arm 1: Hydroxychloroquine Sulfate + Azithromycin | Arm 2: Hydroxychloroquine Sulfate Alone | Arm 3: Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The period of time over which adverse event data was collected is after six days.
Arm/Group | Arm 1: Hydroxychloroquine Sulfate + Azithromycin | Arm 2: Hydroxychloroquine Sulfate Alone | Arm 3: Placebo
All-Cause Mortality (participants affected / at risk) | 4/16 | 4/30 | 1/29
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/30 | 1/29
Other Adverse Events (participants affected / at risk) | 7/16 | 13/30 | 5/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Hydroxychloroquine Sulfate + Azithromycin (N=16) | Arm 2: Hydroxychloroquine Sulfate Alone (N=30) | Arm 3: Placebo (N=29)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Hydroxychloroquine Sulfate + Azithromycin (N=16) | Arm 2: Hydroxychloroquine Sulfate Alone (N=30) | Arm 3: Placebo (N=29)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 6 (8) | 2 (3)
Investigations (Investigations) | 3 (4) | 6 (11) | 2 (2)
Infections and infestations (Infections and infestations) | 1 (2) | 6 (8) | 1 (1)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 2 (3)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT04336332/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT04336332/SAP_001.pdf
  • Informed Consent Form: ICF #1 (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT04336332/ICF_002.pdf
  • Informed Consent Form: ICF #2 (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT04336332/ICF_003.pdf